CLINICAL TRIAL: NCT05638022
Title: Early Detection of Familial Hypercholesterolaemia
Brief Title: Pilot Project of Familial Hypercholesterolemia Screening in Newborns in the Czech Republic
Acronym: CzeCH-IN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: Centre of Cardiovascular and Transplantation Surgery, Czech Republic (Other); The Central European Institute of Technology - Masaryk University (Unknown); Motol University Hospital (Other); Brno University Hospital (Other); Municipal Hospital Ostrava (Other); University Hospital Olomouc (Other); University Hospital Pilsen (Other); Masaryk Hospital in Ústí nad Labem, Regional Health Corporation (Unknown); Regional Hospital Kolín, Hospital of the Central Bohemian Region (Unknown); Havlíčkův Brod Hospital (Unknown); Tomáš Baťa Regional Hospital in Zlín (Unknown); Hospital of Hospitaller Brothers (Unknown); Třebíč Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: UZIS 2021/1
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-06

CONDITIONS: Familial Hypercholesterolaemia
Keywords: Familial Hypercholesterolaemia; Newborns; Screening; Cholesterol; Molecular analysis
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Biospecimen Retention: Samples With DNA — Umbilical Cord blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborns: Newborns matching inclusion criteria
  Interventions: Diagnostic Test: Total cholesterol (TC) level test and direct Low density lipoprotein cholesterol (LDL-C) level test; Diagnostic Test: DNA testing

INTERVENTIONS:
Diagnostic Test: Total cholesterol (TC) level test and direct Low density lipoprotein cholesterol (LDL-C) level test — Total cholesterol (TC) level testing and direct Low density lipoprotein cholesterol (LDL-C) level testing will be performed in all 10,000 newborns enrolled in the project.
Diagnostic Test: DNA testing — DNA testing (NGS analysis of DNA mutations in 9 genes: LDLR, APOB, APOE, PCSK9, LDLRAP1, STAP1, ABCG5, ABCG8, LIPA and polygenic markers) will be performed in the subcohort of 1,500 newborns with highest level of Low density lipoprotein cholesterol (LDL-C).
  Other Names: NGS analysis

SUMMARY:
The project is a national, prospective, multicenter, non-interventional pilot project of screening for the disease Familial hypercholesterolaemia (FH) in newborns in the Czech Republic.

The main goal of the project is to methodically prepare, implement and evaluate a pilot project that will verify the suitability of the proposed procedure of early detection of Familial hypercholesterolaemia in such a way as to ensure the maximum positive impact on the health of the population and high cost-effectiveness of the whole process.

DETAILED DESCRIPTION:
The project is a national, prospective, multicenter, non-interventional pilot project of screening for the disease Familial hypercholesterolaemia in newborns taking place in 12 selected perinatological centers in the Czech Republic. The main goal of the project is to methodically prepare, implement and evaluate a pilot project that will verify the suitability of the proposed procedure of early detection of Familial hypercholesterolaemia in such a way as to ensure the maximum positive impact on the health of the population and high cost-effectiveness of the whole process.

The project will include 10,000 newborns, in whom umbilical cord blood will be taken, from which the level of blood lipids - LDL cholesterol and total cholesterol - will be determined in a biochemical laboratory. In 1,500 newborns with the highest level of LDL cholesterol in the whole examined cohort, a molecular genetic examination of causal DNA mutations responsible for the FH development will be performed. The final evaluation of the FH diagnosis will be performed by specialized doctor, who in case of confirmed/suspected FH diagnosis will contact the child's mother or the pediatrician who has taken the child into care. According to epidemiological data, it can be assumed that the project will newly reveal approximately 40-50 children (families) with FH disease. This approach will allow FH-positive newborns to initiate adequate regimen measures from 2 years of age later followed by pharmacological intervention from 8 years of age, which will dramatically reduce their risk of premature death and non-fatal cardiovascular ischemic events at their young adult age. In addition, according to the valid recommendations for the diagnosis and treatment of this disease in the Czech Republic, it can be assumed that finding FH-positive child will also lead to cascade examination of his/her relatives (parents, grandparents, siblings and possibly also siblings of the affected parent), which, due to the type of FH inheritance, will reveal at least one another FH-positive relative in the affected family. It should be emphasized that the parents of newly diagnosed child are usually at the age when the risk of their untimely death or premature non-fatal myocardial infarction is very high (compared to common population). In adult relatives of the sick child, in whom FH disease will be subsequently diagnosed, the necessary pharmacological treatment will be initiated immediately.

As a result, the pilot project should provide data that will help the relevant authorities to decide on the possible extension of the existing neonatal screening in the Czech Republic to Familial hypercholesterolaemia testing. The project will also raise awareness of Familial hypercholesterolaemia in society.

The project is supported by the European Social Fund (Operational Program Employment) and the state budget of the Czech Republic and is registered by the Ministry of Labour and Social Affairs of the Czech Republic under ID: CZ.03.2.63/0.0/0.0/15_039/0009642.

ELIGIBILITY:
Inclusion Criteria:

1. The mother of the unborn child has a permanent residence in the Czech Republic.
2. The mother of the unborn child is able to understand the information provided in the Informed Consent and in the Consent to the Processing of Personal Data.

Exclusion Criteria:

1. The unborn child suffer from a severe developmental defect. Severe developmental defects are considered to be: severe CNS defect (hydrocephalus, holoprosencephaly), severe heart defect requiring surgical correction, congenital pulmonary airway malformation (CPAM), cystic renal degeneration, GIT obstruction, cleft palate and neural tube defects.
2. The unborn child suffer from growth retardation (premature babies can be included in the project). Growth retardation is considered to be a growth restriction with a weight estimate below the 5th percentile.
3. Either of the future parents (mother / father) is diagnosed with FH (or is aware that he or she would suffer from FH).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any pregnant woman in the Czech Republic (matching inclusion criteria) who will give a birth in one of the 12 perinatological centres participating in the project.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Familial hypercholesterolaemia in screened cohort of newborns | Until December 31, 2022
  Number of newborns with confirmed Familial hypercholesterolaemia in screened cohort based on combination of biochemical and molecular-genetic testing made from umbilical cord blood.
Optimal methodological settings for Familial hypercholesterolaemia detection based on combination of both biochemical and molecular-genetic testing made from umbilical cord blood | Until February 28, 2022
  Optimal settings for Familial hypercholesterolaemia detection from umbilical cord blood: LDL-cholesterol/total cholesterol cut-off values in combination with presence/absence of specific gene mutations/variants.

SECONDARY OUTCOMES:
Up to 10,000 newborns enrolled in the project | Until December 31, 2022
  Up to 10,000 newborns enrolled in the project.

CONTACTS AND LOCATIONS:
Overall Officials: Ondřej Májek, PhD, Principal Investigator — Institute of Health Information and Statistics of the Czech Republic; Tomáš Freiberger, Prof., Study Director — Centre of Cardiovascular and Transplantation Surgery, Czech Republic; Michal Vrablík, Prof., Study Chair — General University Hospital, Prague
Locations (11):
- Czechia (11):
  - Brno University Hospital, Brno
  - Brothers of Charity Hospital, Brno
  - Havlíčkův Brod Hospital, Havlíčkův Brod
  - Regional Hospital Kolín, Hospital of the Central Bohemian Region, Kolín
  - University Hospital Olomouc, Olomouc
  - Municipal Hospital Ostrava, Ostrava
  - University Hospital Pilsen, Pilsen
  - Motol University Hospital, Prague
  - Třebíč Hospital, Třebíč
  - Masaryk Hospital in Ústí nad Labem, Regional Health Corporation, Ústí nad Labem
  - Tomáš Baťa Region Hospital in Zlín, Zlín

IPD SHARING:
Plan to Share IPD: No